CLINICAL TRIAL: NCT01208909
Title: Combined Approach to GBM-resection by 5-ALA and Intraoperative MRI
Brief Title: Combined Approach to Resection of Glioblastoma (GBM) by 5-Aminolevulinic Acid (5-ALA) and Intraoperative Magnetic Resonance Imaging (MRI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Dr. R. L. Bernays, University of Zurich
Other Study IDs: ZU-XYZ-002
Record Dates: First submitted 2010-04-13; First posted 2010-09-24 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tumor samples for pathophysiology
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: diagnostic 5-ALA and MRI for tumor resection — diagnostic 5-ALA and MRI for tumor resection

SUMMARY:
In the treatment of glioblastoma (GBM) neurosurgical resection of the tumor is usually considered a a first step of effective therapy. Radical resection of the tumor is highly beneficial to the patient as measured in progression-free survival and overall survival. At the same time eloquent areas of the brain have to remain intact to preserve quality of life.

Both 5-ALA fluorescence and intraoperative MRI are used for intraoperative marking of tumor tissue and thereby to improve precision of GBM-Resection.

We now study whether the combination of 5-ALA fluorescence and intraoperative MRI increases the number of sites where tumor tissue can be detected.

- Trial with surgical intervention

DETAILED DESCRIPTION:
Precision of GBM-Resection Intraoperative marking of tumor tissue Combination of 5-ALA fluorescence and intraoperative MRI

ELIGIBILITY:
Inclusion criteria:

* patients with Glioblastoma multiforme (GBM)
* no other tumor types or metastases

Exclusion criteria:

* Allergy against 5-ALA or Porphyrin
* Porphyria
* Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Glioblastoma multiforme (GBM)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: René L Bernays, MD, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- UniversitätsSpital Zürich, Zurich, Switzerland